CLINICAL TRIAL: NCT05465707
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation, Multiple-dose Phase Ib/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Efficacy of CM313 Injection in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study of CM313 Injection in Subjects With Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM313-106001
Record Dates: First submitted 2022-07-07; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CM313 2 mg/kg (Experimental): Once 1 week, intravenous infusion.
  Interventions: Biological: CM313 2 mg/kg
- CM313 4 mg/kg (Experimental): Once 1 week, intravenous infusion.
  Interventions: Biological: CM313 4 mg/kg
- CM313 8 mg/kg (Experimental): Once 1 week, intravenous infusion.
  Interventions: Biological: CM313 8 mg/kg
- CM313 16 mg/kg (Experimental): Once 1 week, intravenous infusion.
  Interventions: Biological: CM313 16 mg/kg
- Placebo (Placebo Comparator): Once 1 week, intravenous infusion.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CM313 2 mg/kg — Once 1 week, intravenous infusion.
  Arms: CM313 2 mg/kg
Biological: CM313 4 mg/kg — Once 1 week, intravenous infusion.
  Arms: CM313 4 mg/kg
Biological: CM313 8 mg/kg — Once 1 week, intravenous infusion.
  Arms: CM313 8 mg/kg
Biological: CM313 16 mg/kg — Once 1 week, intravenous infusion.
  Arms: CM313 16 mg/kg
Biological: Placebo — Once 1 week, intravenous infusion.
  Arms: Placebo

SUMMARY:
A study of CM313 in subjects with systemic lupus erythematosus

DETAILED DESCRIPTION:
This is a multi-center, randomed, open-label, dose escalation and dose expansion, Phase 1 study to evaluate the safety, tolerability, Pharmacokinetics and preliminary anti-tumor activity.

About 40 patients who meet eligibility criteria will be randomized 4:1 to receive either CM313 or matched placebo, intravenous infusion.

The treatment period includes single dosing and multiple dosing period, in which CM313 and placebo will be adminitrated intravenously, once every 1 week.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 65 years old.
* Positive autoantibody serology test at screening.
* Contraception.
* Voluntarily sign the ICF.

Exclusion Criteria:

* With central nervous system disease caused by or not caused by SLE within 8 weeks before the first dose of study drug.
* Possibly active Mycobacterium tuberculosis infection.
* With the history of vital organ transplantation or hematopoietic stem cell/or bone marrow transplantation.
* Heavy drinking in the 3 months prior to screening.
* With depression or suicidal thoughts.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs). | Baseline up to Day 113
  Safety parameters

REFERENCES:
- [Derived] Zhao J, Lin C, Xie Q, Shu Q, Cui Y, Luo H, Fan W, Huang A, Zhao Y, Fu Z, Xie C, Wu H, Yang N, He L, Feng P, Zhang T, Zhou H, Liu W, Hou Q, Mao X, Sun J, Chen B, Zeng X. Anti-CD38 monoclonal antibody CM313 for systemic lupus erythematosus: a randomized, double-blind, placebo-controlled phase Ib/IIa trial. Signal Transduct Target Ther. 2025 Nov 26;10(1):383. doi: 10.1038/s41392-025-02487-2. PMID 41290616